CLINICAL TRIAL: NCT06182904
Title: Management of Pilon Fractures With Versus Without Fibula Fixation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Mofdy Shafik kaeen, Resident, Assiut University
Other Study IDs: pilon fractures
Record Dates: First submitted 2023-06-30; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Pilon Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Management of pilon fractures with fibula fixation
  Interventions: Device: Dynamic compression plate
- 2: Management of pilon fracture without fibula fixation

INTERVENTIONS:
Device: Dynamic compression plate — Fixation of fibula in some cases with dynamic compression plate
  Groups: 1

SUMMARY:
Management of pilon fractures with versus without fibula fixation

DETAILED DESCRIPTION:
Comparing results with or without fibular fixation in :

* Rate of bone union .
* Functional return ( clinical outcomes)
* Alignment of lower limb.

ELIGIBILITY:
Inclusion Criteria:

* patients with metaphyseal non rotational pilon or distal tibia : age ( 18 _ 65 )
* No skin troubles
* No infections
* Non-dibetic patients.

Exclusion Criteria:

* Patients who will not complete their follow up.
* Skin troubles
* Infections

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Management of pilon fractures with versus withot fibula fixation: prospective controlled study
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-03-21 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Fracture healing and bone union | Baseline
  by RUST score

SECONDARY OUTCOMES:
Incidece and rate of complications | Baseline
  Incidence and rate of complications (e.g. non-union, skin breakdown , infections and postraumatic malaligment) by AOFAS score